CLINICAL TRIAL: NCT00163605
Title: A Prospective Clinical Study to Evaluate the Performance and Safety of the Bone Substitute MBCP-FS in Maxillary Sinus Lift Procedures
Brief Title: Performance and Safety of Bone Substitute MBCP-FS in Maxillary Sinus Lift Procedures
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 570201
Record Dates: First submitted 2005-09-08; First posted 2005-09-14 (Estimated); Last update posted 2007-11-15 (Estimated); Status verified 2007-11

CONDITIONS: Sinus Implant Reconstruction
Keywords: Sinus augmentation; Alloplastic bone substitute; Hydroxyl apatite

INTERVENTIONS:
Device: Macroporous Biphasic Calcium Phosphate-Fibrin Sealant Vapor Heated Solvent/Detergent Treated 4 IU/ML Thrombin (MBCP-FS)

SUMMARY:
The purpose of this study is to evaluate the performance and to monitor the safety of the bone substitute Macroporous Biphasic Calcium Phosphate-Fibrin Sealant Vapor Heated Solvent/Detergent Treated 4 IU/ML Thrombin (MBCP-FS) in Sinus Lift Procedures . This study will be conducted in two parts: part A evaluates safety and performance of MBCP-FS in bone regeneration i.e. the amount of new bone that is formed and its suitability for dental implant placement. Part B is designed to evaluate long-term safety and performance of the product, i.e. whether the newly-formed bone is suitable to retain implants.

ELIGIBILITY:
Inclusion criteria:

* Written informed consent obtained from the subject prior to participation in the study
* At least 18 years of age
* Partially or totally edentulous with an atrophic posterior maxilla requiring unilateral or bilateral sinus lift before dental implant placement
* In case of bilateral sinus lifts, both sides are operated on the same day.
* Subjects with remaining minimal maxillary bone height between 2 mm and 5 mm at the site with minimal height in the area where implants are planned, and a remaining maxillary bone thickness >= 5 mm in the area where implants are planned

Exclusion Criteria:

* Previous or coeval major surgical intervention in the targeted area, or major surgical intervention in the targeted area planned within the next 18 months (like Caldwell Luc) (minor interventions like surgical tooth extraction or root tip resections are allowed)
* Surgical tooth extraction in the targeted area less than three months before the SLP
* Maxillary and sinus disorders including: acute sinusitis, chronic sinus pathology, retained root tips, polyps, tumors, and cysts in antral cavity or odontogenic cysts, alveolar scar ablation
* Major occlusal disturbance, like severe bruxism
* Uncontrolled* periodontal disease
* An inadequate interarch distance requiring an oppositional graft
* Immune system disorders, immunodeficiency or immunosuppression
* Known coagulation disorder
* Uncontrolled* diabetes mellitus
* Severe hyperparathyroidism
* Receiving long-term anti-inflammatory treatment with NSAIDs or corticosteroids
* Chemotherapy current or in the last three months
* Having undergone maxillary radiation therapy
* Known hypersensitivity to aprotinin or to other components of the investigational product
* Abuse of alcohol or drugs or tobacco consumption of more than 5 cigarettes per day at study start
* Non-compliant for future dental hygiene
* Severely compromised physical and psychological health, that in the investigators opinion will affect patient compliance
* Any contra-indications to the use of MBCP, which are defined as osteomyelitis, degenerative bone disease or necrosis of the recipient site
* Concurrently participating in another clinical trial and having received another investigational drug or device within the last 30 days
* Pregnant or lactating, or intending to become pregnant during the study period

  * Uncontrolled = not treated or not stabilized after treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86
Dates: Start 2004-09; Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Baxter BioScience Investigator, Principal Investigator — Baxter BioScience
Locations (3):
- Germany (3):
  - Klinik für Mund-, Kiefer- und Gesichtschirurgie des Helios-Klinikums Erfurt, Erfurt
  - Klinik und Poliklinik für Mund-, Kiefer- und Gesichtschirurgie der Universität Erlangen-Nürnberg, Erlangen
  - Universitätsklinikum Schleswig Holstein, Campus Kiel, Kiel